CLINICAL TRIAL: NCT01228097
Title: Changes in Neural Response to Eating After Bariatric Surgery: MRI Results
Brief Title: Neural Response to Eating and Weight Status
Acronym: NEWS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: R01DK085615 (NIH)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2011-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be drawn for safety labs. Blood plasma will be archived for analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Gastric Bypass: Participants who receive gastric bypass surgery.
- Principally Restrictive Surgery: Participants who receive gastric banding or sleeve gastrectomy surgery.
- Weight Stable: Participants who remain weight stable.

SUMMARY:
This study will compare brain and hormone responses to food images (and food) in women who undergo: (1) gastric bypass surgery; (2) principally restrictive surgery (laparoscopic adjustable gastric banding or laparoscopic sleeve gastrectomy); or (3) no weight loss surgery, with the intent of remaining relatively weight stable (within 10-15 lb of your present weight). The investigators will use magnetic resonance imaging (MRI) to see how the brain responds to pictures of food and to consuming a liquid meal replacement. The investigators wish to determine whether the two surgeries have different effects on appetite, as observable in the brain, and whether the possible effects on appetite differ from those in participants who have a similar body weight but remain relatively weight stable. The investigators also will draw blood to determine how "hunger" and "fullness" hormones change after eating and to see if there are any differences among the three groups. The study is being sponsored by the National Institutes of Health (NIH).

DETAILED DESCRIPTION:
We hypothesize that RYGB-treated patients will exhibit greater reductions (from baseline) in BOLD response in areas associated with homeostatic and hedonic eating than will both LAGB/LSG and control patients. We also expect that LAGB/LSG patients (as a result of hormonal changes occurring with weight loss) will display greater increases in BOLD response to images of highly palatable foods than will extremely obese controls.

We expect that RYGB-treated patients will show larger increases (relative to baseline) in postprandial GLP-1 and PYY3-36 than the LAGB/LSG and obese control groups. We will also compare changes in ghrelin in the three groups. We predict that patients who undergo RYGB will have greater reductions in ghrelin than will control subjects.

We expect that RYGB-treated patients will demonstrate greater postprandial changes (relative to baseline) in brain activity in the homeostatic and hedonic feeding areas (suggesting normalization of satiety and of neural processing of food reward) than will patients who undergo LAGB/LSG or who do not seek weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Over 18 years old
* BMI of 40 kg/ m2 (or 35 kg/m2 in the presence of significant weight-related comorbidities, including established coronary artery disease, established peripheral arterial disease, symptomatic carotid artery disease, sleep apnea, metabolic syndrome, cardiomyopathy, hypertension, and debilitating joint pain).
* Non-surgical group must be willing to remain weight stable and not seek weight loss (i.e., defined as remaining within 5% of baseline weight).

Exclusion Criteria:

* Weight > 350 pounds the maximum weight that can be accommodated in the scanner); supine abdominal width (with arms folded above) > 60 cm or sagittal diameter > 50 cm (i.e., these are the maximum dimensions that can be accommodated in the scanner)
* Pregnancy or lactation
* Type 1 or type 2 diabetes
* Severe major depression or other psychiatric disorder that significantly interferes with daily living
* Substance use disorder (current or in remission 1 year)
* Current use of nicotine or any illicit drug
* Presence or history of orthopedic circumstances, metallic inserts, pacemaker, claustrophobia, or other conditions that may interfere with magnetic resonance imaging
* Use of weight loss medications or other agents known to affect body weight or blood glucose (e.g., glucocorticoids, second-generation antipsychotic medications)
* Lack of capacity to provide informed consent
* Non-surgical participants interested in losing weight in the next 2 years
* Plans to relocate from the area within 2 years
* Principal Investigator discretion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with extreme obesity (i.e., BMI 40 kg/m2) or moderate obesity (BMI 35.0-39.9 kg/m2) plus significant weight-related comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To compare changes in BOLD response to images of high-calorie foods in RYGB patients, LAGB/LSG patients, and untreated controls. | Baseline, 6-Months, 18-Months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Wadden, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Sarkar S, Anokye-Danso F, Tronieri JS, Millar JS, Alamuddin N, Wadden TA, Ahima RS. Differential Effects of Roux-en-Y Gastric Bypass Surgery and Laparoscopic Sleeve Gastrectomy on Fatty Acid Levels. Obes Surg. 2019 Dec;29(12):3941-3947. doi: 10.1007/s11695-019-04062-5. PMID 31290107
- [Derived] Alamuddin N, Vetter ML, Ahima RS, Hesson L, Ritter S, Minnick A, Faulconbridge LF, Allison KC, Sarwer DB, Chittams J, Williams NN, Hayes MR, Loughead JW, Gur R, Wadden TA. Changes in Fasting and Prandial Gut and Adiposity Hormones Following Vertical Sleeve Gastrectomy or Roux-en-Y-Gastric Bypass: an 18-Month Prospective Study. Obes Surg. 2017 Jun;27(6):1563-1572. doi: 10.1007/s11695-016-2505-5. PMID 28004304